CLINICAL TRIAL: NCT00045916
Title: Optimization of Electroconvulsive Therapy
Brief Title: Optimizing Electroconvulsive Therapy for Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #3891; R01MH061609 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2002-09-13; First posted 2002-09-17 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2008-10

CONDITIONS: Depression; Depressive Disorder; Bipolar Disorder
Keywords: Electroconvulsive therapy; Antidepressive Agents
MeSH Terms: conditions — Depression; Depressive Disorder; Bipolar Disorder | interventions — Nortriptyline; Venlafaxine Hydrochloride; Lithium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- High dosage ECT + nortriptyline (Experimental): Participants will receive nortriptyline and high dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment.
  Interventions: Procedure: High dosage electroconvulsive therapy; Drug: Nortriptyline; Drug: Lithium
- High dosage ECT + venlafaxine (Experimental): Participants will receive venlafaxine and high dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment.
  Interventions: Procedure: High dosage electroconvulsive therapy; Drug: Venlafaxine; Drug: Lithium
- High dosage ECT + placebo (Placebo Comparator): Participants will receive placebo and high dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment weeks.
  Interventions: Procedure: High dosage electroconvulsive therapy; Drug: Lithium
- Low dosage ECT + nortriptyline (Experimental): Participants will receive nortriptyline and high dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment.
  Interventions: Drug: Nortriptyline; Drug: Lithium; Procedure: Low dosage electroconvulsive therapy
- Low dosage ECT + venlafaxine (Experimental): Participants will receive venlafaxine and low dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment.
  Interventions: Drug: Venlafaxine; Drug: Lithium; Procedure: Low dosage electroconvulsive therapy
- Low dosage ECT + placebo (Experimental): Participants will receive placebo and low dosage ECT. If the ECT is effective participants will receive lithium after ECT treatment weeks.
  Interventions: Drug: Lithium; Procedure: Low dosage electroconvulsive therapy

INTERVENTIONS:
Procedure: High dosage electroconvulsive therapy — Participants will receive high dosage right unilateral ECT at six times the seizure threshold.
  Arms: High dosage ECT + nortriptyline; High dosage ECT + placebo; High dosage ECT + venlafaxine
Drug: Nortriptyline — Participants will receive nortriptyline.
  Arms: High dosage ECT + nortriptyline; Low dosage ECT + nortriptyline
Drug: Venlafaxine — Participants will receive venlafaxine.
  Arms: High dosage ECT + venlafaxine; Low dosage ECT + venlafaxine
Drug: Lithium — Participants will receive lithium.
Procedure: Low dosage electroconvulsive therapy — Participants will receive low dosage bilateral ECT at one and a half times the seizure threshold.
  Arms: Low dosage ECT + nortriptyline; Low dosage ECT + placebo; Low dosage ECT + venlafaxine

SUMMARY:
This study will evaluate the effectiveness of electroconvulsive therapy (ECT) administered with medication for the treatment of a major depressive episode (unipolar or bipolar) and will compare two types of ECT.

DETAILED DESCRIPTION:
This study addresses 2 issues in the optimization of ECT in patients with major depression: whether patients treated with ECT should receive concurrent treatment with antidepressant medications, and the relative efficacy and side effects of high dosage right unilateral (RUL) ECT compared to low dosage bilateral (BL) ECT.

This study has 2 phases. In Phase I, patients are randomized to receive nortriptyline, venlafaxine (Effexor), or placebo while they simultaneously receive either high dosage RUL ECT or low dosage BL ECT. Patients have an electrocardiogram (EKG), a chest x-ray, medical and neurological examinations, and blood tests. Memory function is assessed before and after ECT. Whenever feasible, patients are withdrawn from all prior psychotropic medication before the start of ECT. ECT is administered 3 times per week to inpatients and twice a week to outpatients. Patients continue ECT until they are asymptomatic or until there is a plateau in improvement over 2 treatments.

Patients who respond to ECT enter Phase II and add lithium to either nortriptyline or venlafaxine within 1-3 days of the last ECT. Clinical and side effect evaluations and blood level determinations are conducted weekly for the first month, every 2 weeks until Week 12, and every 4 weeks for the remaining 12 weeks. Following any indication of relapse, patients are monitored more intensively and are re-evaluated within 1 week. The neurocognitive battery is readministered to all patients at 2 and 6 months after the acute ECT course, regardless of ECT clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode (unipolar or bipolar)
* Pre-ECT score of 20 or higher on Hamilton Rating Scale for Depression
* Able to withdraw psychotropic drugs (up to 3 mg/day lorazepam allowed)
* ECT indicated

Exclusion Criteria:

* Schizophrenia, schizoaffective disorder, or other psychosis
* Amnestic disorder, dementia, or delirium
* Pregnancy
* Epilepsy
* Current alcohol or substance abuse or dependence
* CNS disease or brain injury not associated with psychotropic drug exposure
* ECT in the past 6 months
* Medical contraindication for treatment with either nortriptyline or venlafaxine, including allergy to amitriptyline, nortriptyline, or venlafaxine; narrow angle glaucoma; sinus node disease; bundle branch disease; myocardial infarction; coronary artery bypass or angioplasty; or angina
* Type I antiarrhythmic medication
* Supine blood pressure >= 170 mmHg systolic or >= 105 mmHg diastolic at 3 readings over 2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2001-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive battery | Measured at baseline and at 2 and 6 months after the acute ECT course
Clinical evaluations, side effect evaluations, and blood level determinations | Measured weekly for the first month, every 2 weeks until Week 12, and every 4 weeks for the remaining 12 weeks

SECONDARY OUTCOMES:
Memory function | Measured before and after ECT

CONTACTS AND LOCATIONS:
Overall Officials: Harold A. Sackeim, PhD, Study Chair — New York State Psychiatric Institute and Columbia University
Locations (4):
- United States (4):
  - Washington University, St Louis, Missouri
  - New York State Psychiatric Institute at Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Sackeim HA, Haskett RF, Mulsant BH, Thase ME, Mann JJ, Pettinati HM, Greenberg RM, Crowe RR, Cooper TB, Prudic J. Continuation pharmacotherapy in the prevention of relapse following electroconvulsive therapy: a randomized controlled trial. JAMA. 2001 Mar 14;285(10):1299-307. doi: 10.1001/jama.285.10.1299. PMID 11255384
- [Background] Sackeim HA, Prudic J, Devanand DP, Nobler MS, Lisanby SH, Peyser S, Fitzsimons L, Moody BJ, Clark J. A prospective, randomized, double-blind comparison of bilateral and right unilateral electroconvulsive therapy at different stimulus intensities. Arch Gen Psychiatry. 2000 May;57(5):425-34. doi: 10.1001/archpsyc.57.5.425. PMID 10807482
- [Background] McCall WV, Reboussin DM, Weiner RD, Sackeim HA. Titrated moderately suprathreshold vs fixed high-dose right unilateral electroconvulsive therapy: acute antidepressant and cognitive effects. Arch Gen Psychiatry. 2000 May;57(5):438-44. doi: 10.1001/archpsyc.57.5.438. PMID 10807483
- [Derived] McCall WV, Reboussin D, Prudic J, Haskett RF, Isenberg K, Olfson M, Rosenquist PB, Sackeim HA. Poor health-related quality of life prior to ECT in depressed patients normalizes with sustained remission after ECT. J Affect Disord. 2013 May;147(1-3):107-11. doi: 10.1016/j.jad.2012.10.018. Epub 2012 Nov 15. PMID 23158959